CLINICAL TRIAL: NCT02542930
Title: A Phase II Study of Radiotherapy and ZADAXIN's® (Thymalfasin) Induced Abscopal Effect in Patients With Heavily Pretreated, Metastatic Non-small Cell Lung Cancer.
Brief Title: Abscopal Effect for Metastatic Non-small Cell Lung Cancer.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No recruitment.
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Min Fang, MD, Zhejiang Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Zhejiang Provincal People's Hp
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Non-small Cell Lung Cancer; Metastatic Non-small Cell Lung Cancer; Radiotherapy; Thymalfasin
Keywords: Non-small cell lung cancer; Metastatic Non-small cell lung cancer; Radiotherapy; Thymalfasin; ZADAXIN's®
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy; Thymalfasin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiotherapy and Thymalfasin arm (Experimental): Patients with metastatic lesions of Non-small cell lung cancer receiving 3.5Gy per fraction to a total dose of 35Gy/10 fractions over 2 weeks with concurrent thymalfasin;
  Interventions: Radiation: Radiotherapy; Drug: Thymalfasin

INTERVENTIONS:
Radiation: Radiotherapy — Metastatic lesions of Non-small cell lung cancer receiving 3.5Gy per fraction to a total dose of 35Gy/10 fractions over 2 weeks with concurrent thymalfasin.
Drug: Thymalfasin — Metastatic lesions of Non-small cell lung cancer receiving 3.5Gy per fraction to a total dose of 35Gy/10 fractions over 2 weeks with concurrent thymalfasin; Thymalfasin treatment is given twice a week with an interval of 3-4 days each week.
  Other Names: ZADAXIN's®

SUMMARY:
Patients with Non-small cell lung cancer that had metastatic lesions after been treated with definitive surgery or chemoradiotherapy are being asked to participate in this study.

1. To observe immunity-mediated tumor response outside the radiation field (abscopal effect) after chemoradiotherapy of a metastatic site in metastatic Non-small cell lung cancer patients.
2. To induce the efficacy (effectiveness) of a new combination of therapy, chemoradiotherapy and thymalfasin for heavily pretreated, metastatic Non-small cell lung cancer patients;
3. To explore the role of PET/CT scanning to assess tumor response/abscopal effect.

This study will help find out what abscopal effects (good or bad) the combination of radiotherapy and thymalfasin has on metastatic Non-small cell lung cancer.

DETAILED DESCRIPTION:
1. To observe immunity-mediated tumor response outside the radiation field (abscopal effect) after chemoradiotherapy of a metastatic site in metastatic Non-small cell lung cancer patients.
2. To induce the efficacy (effectiveness) of a new combination of therapy, chemoradiotherapy and thymalfasin for heavily pretreated, metastatic Non-small cell lung cancer patients;
3. To explore the role of PET/CT scanning to assess tumor response/abscopal effect.

Eligible are patients with metastatic Non-small cell lung cancer who have achieved stable disease or have disease progression after systemic therapy (surgery or definitive chemoradiotherapy) and have at least three separate measurable sites of metastatic lesions. Extent of metastatic disease is recorded both at CT and PET/CT scanning. Radiation is given during combined therapy to one of the lesions, 35Gy in 10 fractions over a two week interval, conformally to maximally spare normal tissue or organ. Thymalfasin treatment is given twice a week with an interval of 3-4 days each week. At day 22 radiation is re-started and the same radiation dose is delivered to a second metastatic site, again with thymalfasin. Abscopal response is evaluated by assessing clinical and PET/CT response in the non-irradiated measurable metastatic sites. A Phase II clinical trial based on an optimum two-stage Phase II Simon design is used to conduct this pilot study. Ten patients will be treated in Stage one; if there are no abscopal responses, the trial will be terminated. If there are one or more abscopal responses in Stage One, the trial will proceed to enroll an additional 19 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed colorectal cancer which is persistent and metastatic or recurrent and metastatic;
2. Patients must have at least 3 distinct measurable metastatic sites at least 1 cm of larger in their largest diameter;
3. Age ≥18 years;
4. Metastatic disease measurable on a CT/MRI scan. The primary tumor is not considered measurable disease. Metastatic lesions within a prior radiation field are acceptable as long as disease has progressed in the radiation field by RECIST criteria. The same imaging modality performed at baseline (CT or MRI) will be repeated at subsequent imaging.
5. ECOG performance status: 0-1;
6. Life expectancy ≥ 3 months.
7. Patients have adequate baseline organ and marrow function as defined by an absolute neutrophil count greater than 1500 cells per μL, platelet concentration of greater than 50 000 per μL, total bilirubin less than 1•5 times the upper limit of normal (ULN), aspartate aminotransferase and alanine aminotransferase less than 2•5 times the ULN, and serum creatinine less than 1•5 times the ULN;
8. Signed consent forms voluntarily;

Exclusion Criteria:

1. Patients who have had prior allergic reaction to Apatinib;
2. Patients undergoing therapy with other investigational agents.
3. Women who are pregnant or breastfeeding;
4. Patients with known brain metastases can be included in this clinical trial but brain lesions are not eligible as target or non target lesion;
5. Anticipated patient survival under 3 months;
6. Active severe infection or known chronic infection with HIV, hepatitis B virus, or hepatitis C virus;
7. Cardiovascular disease problems including unstable angina, therapy for life-threatening ventricular arrhythmia, myocardial infarction, stroke or congestive heart failure within the last 6 months;
8. The subject has had another active malignancy within the past five years except for cervical cancer in site, in situ carcinoma of the bladder or non-melanoma carcinoma of the skin;
9. Clinically significant and uncontrolled major medical conditions including but not limited to: active uncontrolled infection, symptomatic congestive heart failure, Unstable angina pectoris or cardiac arrhythmia, psychiatric illness/ social situation that would limit compliance with study requirements; any medical condition, which in the opinion of the study investigator places the subject at an unacceptably high risk for toxicities;
10. Patients with any other concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for participation in the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with an abscopal response assessed at 7-8 weeks after the initiation of treatment. | week 7- week 8

SECONDARY OUTCOMES:
The number of participants with adverse events from the date of enrollment until 2 years from the opening of the study. | year 0- year 2
The proportion of patients alive with abscopal responses from the date of enrollment until date of death from any cause, assessed up to 2 years from the opening of the study. | year 0- year 2

CONTACTS AND LOCATIONS:
Overall Officials: Shuqiang Wu, MD, Study Chair — Zhejiang Provincial People's Hospital; Yongshi Jia, MD, Study Chair — Zhejiang Provincial People's Hospital

REFERENCES:
- [Background] Golden EB, Chhabra A, Chachoua A, Adams S, Donach M, Fenton-Kerimian M, Friedman K, Ponzo F, Babb JS, Goldberg J, Demaria S, Formenti SC. Local radiotherapy and granulocyte-macrophage colony-stimulating factor to generate abscopal responses in patients with metastatic solid tumours: a proof-of-principle trial. Lancet Oncol. 2015 Jul;16(7):795-803. doi: 10.1016/S1470-2045(15)00054-6. Epub 2015 Jun 18. PMID 26095785